CLINICAL TRIAL: NCT00331344
Title: Phase I/II Trial of Epothilone Analog BMS-247550 (Ixabepilone), Mitoxantrone, and Prednisone in Hormone Refractory Prostate Cancer (HRPC) Patients Previously Treated With Chemotherapy
Brief Title: Treating Patients With Metastatic Prostate Cancer Not Responding to Hormone and Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00155; 055513; CDR0000481121 (Registry Identifier: PDQ (Physician Data Query)); N01CM62202 (NIH); NCT01648374 (obsolete NCT alias)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mitoxantrone; ixabepilone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive mitoxantrone hydrochloride IV over 30 minutes and ixabepilone IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: mitoxantrone hydrochloride; Drug: ixabepilone; Drug: prednisone

INTERVENTIONS:
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra

SUMMARY:
This phase I/II trial is studying the side effects and best dose of ixabepilone and mitoxantrone hydrochloride when given together with prednisone and to see how well they work in treating patients with metastatic prostate cancer that did not respond to hormone therapy and chemotherapy. Drugs used in chemotherapy, such as ixabepilone, mitoxantrone hydrochloride, and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and dose-limiting toxicities of the combination of ixabepilone, mitoxantrone hydrochloride, and prednisone in patients with hormone-refractory metastatic prostate cancer that progressed during or after taxane-based chemotherapy. (Phase I) II. Assess the efficacy, as measured by reduction in prostate-specific antigen, of this regimen in these patients. (Phase II)

SECONDARY OBJECTIVES:

I. Evaluate the overall safety of this regimen as second-line chemotherapy in these patients.

II. Evaluate the objective response rate in patients treated with this regimen.

OUTLINE: This is a multicenter, phase I, open label, dose-escalation study of mitoxantrone hydrochloride and ixabepilone followed by a phase II study.

PHASE I: Patients receive mitoxantrone hydrochloride intravenously (IV) over 30 minutes and ixabepilone IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of mitoxantrone hydrochloride and ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive mitoxantrone hydrochloride and ixabepilone at the MTD determined in phase I and prednisone as in phase I.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Progressive metastatic disease (i.e., positive bone scan or measurable disease) despite castrate levels of testosterone (either from orchiectomy or luteinizing hormone-releasing hormone [LHRH] agonist therapy)

  * Progressive disease after discontinuing hormonal therapy
  * Progressive disease is based on any of the following*:

    * Transaxial imaging
    * Rise in prostate-specific antigen (PSA)
    * Radionuclide bone scan (must show new metastatic lesions)
* Nonmeasurable or measurable disease

  * For measurable disease, progression is defined by RECIST criteria
  * Positive bone scan and elevated PSA required for nonmeasurable disease

    * PSA evidence of progressive prostate cancer during or after first-line chemotherapy consists of a PSA level ≥ 2 ng/mL that has risen on ≥ 2 successive occasions ≥ 1 week apart
* Received ≥ 3 prior courses of paclitaxel- or docetaxel-based therapy, with disease progression documented during therapy or after cessation of therapy

  * No more than 1 prior chemotherapy regimen
  * Re-treatment with the same taxane-based regimen allowed
  * Changes in prior chemotherapy regimen (addition of other agents) for disease progression are considered 2 chemotherapy regimens, and are not allowed
* PSA ≥ 2 ng/mL
* Testosterone < 50 ng/dL

  * Patients must continue primary androgen deprivation with LHRH analogue if they have not undergone orchiectomy
* No known active brain metastases
* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance > 40 mL/min
* ALT and AST < 2.5 times ULN
* Granulocyte count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin < 1.5 times ULN
* Ejection fraction normal by MUGA scan or echocardiogram
* No significant cardiovascular disease, including any of the following:

  * Congestive heart failure (New York Heart Association class III-IV heart disease)
  * Active angina pectoris
  * Myocardial infarction within the past 6 months
* No serious infections or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by study therapy
* No psychiatric illness or social situation that would preclude study compliance
* No pre-existing motor or sensory peripheral neuropathy > grade 1
* No known prior severe hypersensitivity reactions to agents containing Cremophor® EL
* No "currently active" second malignancy other than nonmelanoma skin cancer

  * Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered to be at < 30% risk of relapse
* Fertile patients must use effective contraception prior to, during, and for 3 months after completion of study treatment
* See Disease Characteristics
* No prior mitoxantrone hydrochloride, ixabepilone, or other epothilones
* At least 4 weeks since prior hormonal therapy (i.e., any dose of megestrol, finasteride, or any herbal product known to decrease PSA levels [e.g., saw palmetto or PC-SPES]) other than LHRH agonist or a stable dose of corticosteroids from a prior chemotherapy regimen
* More than 4 weeks since other prior systemic therapies for prostate cancer
* At least 4 weeks since prior radiation therapy
* More than 8 weeks since prior radiopharmaceuticals (e.g., strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium)
* No concurrent moderate to strong CYP3A4 inhibitors
* No concurrent prophylactic colony-stimulating factors
* No concurrent radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Harzstark, Principal Investigator — University of California San Francisco Medical Center-Mount Zion
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Result] Rosenberg JE, Ryan CJ, Weinberg VK, Smith DC, Hussain M, Beer TM, Ryan CW, Mathew P, Pagliaro LC, Harzstark AL, Sharib J, Small EJ. Phase I study of ixabepilone, mitoxantrone, and prednisone in patients with metastatic castration-resistant prostate cancer previously treated with docetaxel-based therapy: a study of the department of defense prostate cancer clinical trials consortium. J Clin Oncol. 2009 Jun 10;27(17):2772-8. doi: 10.1200/JCO.2008.19.8002. Epub 2009 Apr 6. PMID 19349545
- [Result] Harzstark AL, Rosenberg JE, Weinberg VK, Sharib J, Ryan CJ, Smith DC, Pagliaro LC, Beer TM, Liu G, Small EJ. Ixabepilone, mitoxantrone, and prednisone for metastatic castration-resistant prostate cancer after docetaxel-based therapy: a phase 2 study of the Department Of Defense Prostate Cancer Clinical Trials Consortium. Cancer. 2011 Jun 1;117(11):2419-25. doi: 10.1002/cncr.25810. Epub 2010 Dec 29. PMID 24048789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (incl. currently followed in these practices, as well as those referred from outside providers) will be screened for interest and eligibility by medical oncologists from UCSF Urologic Oncology Practice CCC, UCSF-VA Medical Cntr, OHSU Cancer Inst., MD Anderson Cancer Cntr, UMich Comprehensive Cancer Cntr and the Portland VA Medical Cntr.
Groups:
- Phase I Group I: Patients receive mitoxantrone hydrochloride 8mg/m2 IV over 30 minutes and ixabepilone 20mg/m2 IV over 3 hours on day 1 and oral prednisone 5mg twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group II: Patients receive mitoxantrone hydrochloride 8mg/m2 IV over 30 minutes and ixabepilone 25mg/m2 IV over 3 hours on day 1 and oral prednisone 5mg twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group III: Patients receive mitoxantrone hydrochloride 10mg/m2 IV over 30 minutes and ixabepilone 25mg/m2 IV over 3 hours on day 1 and oral prednisone 5mg twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group IV: Patients receive mitoxantrone hydrochloride 10mg/m2 IV over 30 minutes and ixabepilone 30mg/m2 IV over 3 hours on day 1 and oral prednisone 5mg twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group V: Patients receive mitoxantrone hydrochloride 12mg/m2 IV over 30 minutes and ixabepilone 30mg/m2 IV over 3 hours on day 1 and oral prednisone 5mg twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group VI: Patients receive mitoxantrone hydrochloride 12mg/m2 IV over 30 minutes and ixabepilone 35mg/m2 IV over 3 hours on day 1 and oral prednisone 5mg twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group Va; Phase II: Patients receive mitoxantrone hydrochloride 12mg/m2 IV over 30 minutes and ixabepilone 30mg/m2 IV over 3 hours on day 1 and pegfilgrastim 6mg SC on day 2 and oral prednisone 5mg twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  pegfilgrastim: Given SC
  prednisone: Given orally
- Phase I Group VIa: Patients receive mitoxantrone hydrochloride 12mg/m2 IV over 30 minutes and ixabepilone 35mg/m2 IV over 3 hours on day 1 and pegfilgrastim 6mg SC on day 2 and oral prednisone 5mg twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  pegfilgrastim: Given SC
  prednisone: Given orally
Period: Phase I
Arm/Group | Phase I Group I | Phase I Group II | Phase I Group III | Phase I Group IV | Phase I Group V | Phase I Group VI | Phase I Group Va | Phase I Group VIa | Phase II
Started | 3 | 3 | 3 | 6 | 6 | 5 | 4 | 6 (1 participant who was enrolled died prior to initiating protocol therapy.) | 0
Completed | 3 | 3 | 3 | 5 (1 participant reached dose limiting toxicity) | 4 (2 participants reached dose limiting toxicity) | 3 (2 participants reached dose limiting toxicity) | 4 | 5 (1 participant reached dose limiting toxicity) | 0
Not Completed | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0
Period: Phase II
Arm/Group | Phase I Group I | Phase I Group II | Phase I Group III | Phase I Group IV | Phase I Group V | Phase I Group VI | Phase I Group Va | Phase I Group VIa | Phase II
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (6 patients in Phase I Group VIa continued to the Phase II period.) | 52 (Protocol enrollment (63) minus 11 ineligible prior to receiving treatment.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 48
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 50
Age, Continuous [Median (Full Range); unit: years] | 66.7 [39 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 88
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88

OUTCOME MEASURES:

1. Primary Outcome: Proportion Responding to Treatment With of the Combination of Ixabepilone and Mitoxantrone Hydrochloride With Prednisone in Hormone Refractory Prostate Cancer Patients Who Have Had Prior Taxane Chemotherapy Based Upon a PSA Decline of > 50% (Phase II)
Description: Descriptive statistics will be calculated to characterize the disease and treatment factors including the proportion responding with a 95% confidence interval. If accrual is completed and more than 15 of 58 patients show > 50% Prostate Specific Antigen (PSA) declines after 3 courses, then the null hypothesis of a 20% response proportion will be rejected. PSA declines for individual patients will be plotted in the form of a waterfall diagram of maximal PSA declines.
  58 patients were enrolled for phase II, two were ineligible so 56 patients were analyzed.
Time Frame: Every 3 courses until cancer progression/excessive toxicity or death
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Combination Chemotherapy): Patients receive mitoxantrone hydrochloride 12mg/m2 IV over 30 minutes and ixabepilone 35mg/m2 IV over 3 hours on day 1 and pegfilgrastim 6mg SC on day 2 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  pegfilgrastim: Given SC
  prednisone: Given orally
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 56
Participants | 25

2. Primary Outcome: Safety of the Combination of Ixabepilone, Mitoxantrone Hydrochloride, and Prednisone in Patients With Hormone-refractory Metastatic Prostate Cancer That Progressed During or After Taxane-based Chemotherapy (Phase I)
Description: This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 for adverse event monitoring and reporting. The cumulative grade 3 or higher adverse events for all dose levels are noted below and in the table of adverse events.
Time Frame: Every 21 days until cancer progression/excessive toxicity or death
Population: Phase I dose escalation study participants
Measure: Number; unit: Adverse Events (above threshold)
Groups:
- Phase I Treatment (Groups I-VIa): Patients receive mitoxantrone hydrochloride 8-12mg/m2 IV over 30 minutes and ixabepilone 20-35mg/m2 IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Patients in groups Va and VIa also received pegfilgrastim 6mg SC on day 2. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  pegfilgrastim: Given SC
  prednisone: Given orally
Arm/Group | Phase I Treatment (Groups I-VIa)
Number analyzed (Participants) | 36
Adverse Events (above threshold) | 62

3. Primary Outcome: Dose Limiting Toxicities for Each Dose Level of Ixabepilone, Mitoxantrone Hydrochloride, and Prednisone in Patients With Hormone-refractory Metastatic Prostate Cancer That Progressed During or After Taxane-based Chemotherapy (Phase I).
Description: Cohorts of 3 patients will be enrolled at each dose level; if 1 dose limiting toxicity (DLT) is observed then the cohort will be expanded to 6 patients. If a second DLT is observed, the previous dose level will be considered the maximum tolerated dose (MTD). If all observed DLT are due to neuropathy (specific to ixabepilone), then we would consider the previous dose level of Ixabepilone the MTD for that drug, and escalate mitoxantrone hydrochloride as described above to a maximum dose of 12 mg/m^2. Toxicities will be tabulated by grade for each dose cohort and overall for all patients accrued to the phase I study.
Time Frame: Course 1 (first 21 days)
Population: Dose escalation safety study (Phase I)
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Group I: Patients receive mitoxantrone hydrochloride 8 mg/m2 IV over 30 minutes and ixabepilone 20mg/m2 IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase Group II: Patients receive mitoxantrone hydrochloride 8 mg/m2 IV over 30 minutes and ixabepilone 25mg/m2 IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group III: Patients receive mitoxantrone hydrochloride 10 mg/m2 IV over 30 minutes and ixabepilone 25 mg/m2 IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group IV: Patients receive mitoxantrone hydrochloride 10 mg/m2 IV over 30 minutes and ixabepilone 30mg/m2 IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group V: Patients receive mitoxantrone hydrochloride 12 mg/m2 IV over 30 minutes and ixabepilone 30mg/m2 IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group VI: Patients receive mitoxantrone hydrochloride 12 mg/m2 IV over 30 minutes and ixabepilone 35mg/m2 IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  prednisone: Given orally
- Phase I Group Va: Patients receive mitoxantrone hydrochloride 12 mg/m2 IV over 30 minutes and ixabepilone 30mg/m2 IV over 3 hours on day 1 and pegfilgrastim 6mg SC on day 2 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  pegfilgrastim: Given SC
  prednisone: Given orally
- Phase I Group VIa: Patients receive mitoxantrone hydrochloride 12 mg/m2 IV over 30 minutes and ixabepilone 35mg/m2 IV over 3 hours on day 1 and pegfilgrastim 6mg SC on day 2 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  pegfilgrastim: Given SC
  prednisone: Given orally
Arm/Group | Phase I Group I | Phase Group II | Phase I Group III | Phase I Group IV | Phase I Group V | Phase I Group VI | Phase I Group Va | Phase I Group VIa
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 5 | 4 | 6
Participants | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1
Statistical Analysis 1: Comparison: Phase I Group I vs Phase I Group III vs Phase I Group IV vs Phase I Group V vs Phase I Group VI vs Phase I Group Va vs Phase I Group VIa; Cohorts of 3 patients will be enrolled at each dose level; if 1 dose limiting toxicity (DLT) is observed then the cohort will be expanded to 6 patients. If a second DLT is observed, the previous dose level will be considered the MTD. If all observed DLT are due to neuropathy (specific to ixabepilone), then we would consider the previous dose level of Ixabepilone the MTD for that drug, and escalate mitoxantrone hydrochloride as described above to a maximum dose of 12 mg/m^2; Test type: Other; Dose Level VIa = 1 — Dose level VIa (mitoxantrone hydrochloride 12 mg/m2 IV over 30 minutes, ixabepilone 30mg/m2 IV over 3 hours on day 1, pegfilgrastim 6mg SC on day 2, oral prednisone twice daily on days 1-21) was determined to be MTD, based on 1 event of DLT at VIa

4. Secondary Outcome: Time to Progression (Phase II)
Description: Measured from the start of protocol therapy until RECIST (Response Evaluation Criteria In Solid Tumors Criteria) v1.0 progression. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Every 3 months until cancer progression/excessive toxicity or death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 56
months | 4.4 [3.5 to 5.6]

ADVERSE EVENTS:
Groups:
- Phase I and Phase II (Cumulative): Patients in the Phase I period receive mitoxantrone hydrochloride 8-12mg/m2 IV over 30 minutes and ixabepilone 20-35mg/m2 IV over 3 hours on day 1 and oral prednisone twice daily on days 1-21. Patients in groups Va and VIa also received pegfilgrastim 6mg SC on day 2. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients in Phase II receive mitoxantrone hydrochloride 12mg/m2 IV over 30 minutes and ixabepilone 35mg/m2 IV over 3 hours on day 1 and pegfilgrastim 6mg SC on day 2 and oral prednisone twice daily on days 1-21. Treatment repeats every 21 days for ≥ 3 courses in the absence of disease progression or unacceptable toxicity.
  Adverse Events below are reported cumulatively for the entire study.
  mitoxantrone hydrochloride: Given IV
  ixabepilone: Given IV
  pegfilgrastim: Given SC
  prednisone: Given orally
Arm/Group | Phase I and Phase II (Cumulative)
All-Cause Mortality (participants affected / at risk) | 29/88
Serious Adverse Events (participants affected / at risk) | 19/88
Other Adverse Events (participants affected / at risk) | 56/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I and Phase II (Cumulative) (N=88)
Adrenal Insuffiency (Endocrine disorders) | 3
Atrial fibrillation (Cardiac disorders) | 3
Cardiac ischemia/infarction (Cardiac disorders) | 2
Glucose intolerance (Endocrine disorders) | 1
Infection (Prostate) (Renal and urinary disorders) | 1
Infection (limb) (Infections and infestations) | 1
Renal Failure (Metabolism and nutrition disorders) | 2
Pneumonia (Infections and infestations) | 1
Sepsis (Renal and urinary disorders) | 1
Vasovagal episode (Cardiac disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Methicillin-resistant Staphylococcus aureus (Infections and infestations) | 1
Leucocytes (Blood and lymphatic system disorders) | 3
Neutrophil count decreased (Blood and lymphatic system disorders) | 4
Platelet count decreased (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I and Phase II (Cumulative) (N=88)
Hemoglobin (Blood and lymphatic system disorders) | 4
Leucocytes (Blood and lymphatic system disorders) | 17
Lymphopenia (Blood and lymphatic system disorders) | 20
Neutrophil count decreased (Blood and lymphatic system disorders) | 12
Platelet count decreased (Blood and lymphatic system disorders) | 9
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1
Allergic Reaction (Immune system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 8
Atrial tachycardia (Cardiac disorders) | 1
Fatigue (General disorders) | 16
Nausea (Gastrointestinal disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 13
Dizziness (Nervous system disorders) | 2
Dehydration (Gastrointestinal disorders) | 2
Infection, Colon (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Infection, Skin (Infections and infestations) | 4
Pain, Chest (Respiratory, thoracic and mediastinal disorders) | 3
Pain, other (General disorders) | 2
Pain, hip (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (General disorders) | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pain, bone (Musculoskeletal and connective tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Edema, limb (Blood and lymphatic system disorders) | 1
Fever (Infections and infestations) | 1
Hot Flashes (Endocrine disorders) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Peripheral Motor Neuropathy (Nervous system disorders) | 2
Phlebitis (Infections and infestations) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
Taste Alteration (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Weight Loss (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less